CLINICAL TRIAL: NCT04504461
Title: Ambulatory Laparoscopic Inguinal Hernioplasty: Feasibility and Cost Minimization Analysis in a South American Hospital
Brief Title: Ambulatory Laparoscopic Inguinal Hernioplasty: Feasibility and Cost Analysis
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Sponsor
Other Study IDs: 5614
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-08

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Costs and Cost Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laparoscopic Inguinal Hernioplasty. Ambulatory: Laparoscopic Inguinal Hernioplasty performed in ambulatory surgery center
  Interventions: Other: Analysis of feasibility and costs
- Laparoscopic Inguinal Hernioplasty. Hospital Stay: Laparoscopic Inguinal Hernioplasty that have to stay at least 24 hours at the hospital
  Interventions: Other: Analysis of feasibility and costs

INTERVENTIONS:
Other: Analysis of feasibility and costs — Analyze the feasibility and costs of performing laparoscopic inguinal hernioplasty in an ambulatory surgery center

SUMMARY:
Laparoscopic inguinal hernia repair has become one of the elective techniques, attributing the advantages of minimally invasive procedures to it. However, the high costs related to the need for hospitalization and materials make them a limitation at the time of its indication.

The objective is to evaluate the feasibility of performing this procedure in an outpatient surgery center and the cost analysis of an outpatient procedure regarding the same in the setting of hospitalization.

DETAILED DESCRIPTION:
A retrospective analysis was performed on a prospective database in which all patients older than 18 years were included, in which a laparoscopic inguinal hernioplasty was performed in the period between August 2015 and June 2018 in the unit of ambulatory surgery of the Hospital Italiano de Buenos Aires. The same corresponds to an autonomous unit controlled by a health facility with hospitalization, as established by the Asociación Argentina de Cirugía in the Organization Guide and procedures in Ambulatory Surgery.

Laparoscopic repair using a transabdominal preperitoneal technique (TAPP) was proposed for patients with a clinical diagnosis of bilateral inguinal hernia or a recurrent unilateral hernia operated primarily through the anterior approach following the indications for laparoscopic surgery proposed by the European Hernia Society

The demographic data of the patients considered for this study were: age, gender, body mass index (BMI), anesthetic risk according to ASA (American Society of Anesthesiologists) score, comorbidities, bilateral primary or unilateral recurrent hernia, history of previous abdominal surgeries and associated midline hernias The details of the surgical procedure and the ambulatory surgery regimen, as well as possible postoperative complications, were explained to all patients in the preoperative consultation and an informed consent was signed.

The anesthetic technique was the same for everyone. The patients were operated under general anesthesia. Anesthetic induction was performed with propofol 2 mg / kg EV and fentanyl 2 ug / kg EV. Rocuronium 0.6 mg / kg EV was used to facilitate laryngeal mask placement. The anesthetic level was maintained with air, oxygen, sevoflorane at 1.5% expired and with remifentanil (0.25 at 0.5 ug / kg / min) based on the demand of the patient's plan. It was ventilated mechanically in controlled mode. As intraoperative analgesia, ketorolac 1 mg / kg according to renal function or diclofenac 1 mg / kg was used in patients with a history of bronchospasm. This was associated with 8 mg of dexamethasone. Antibiotic prophylaxis during anesthetic induction was performed with cefazolin 2 gr / kg EV.

In 100% of the cases, the surgical technique used was TAPP. The patient was asked to urinate prior to the transfer to the operating room to avoid the placement of a urinary catheter.

With the patient in the supine position, pneumoperitoneum was performed by umbilical scar with closed Veress needle technique. The abdomen was insufflated with a pressure of 12 mmHg. A 10-mm trocar was placed at the umbilical level and two 5-mm trocars were placed on both flanks outside the rectus sheath. In the event that the patient presents with an associated midline hernia, optic trocar was inserted due to hernia defect. It was approached first on one side and then on the contralateral side. After the opening of the peritoneum, dissection of the preperitoneal space and reduction of the hernial content, a polypropylene mesh (Prolene®, Ethicon Johnson & Johnson) of 15 x 12 centimeters was placed covering the myopectineal orifice from the symphysis pubis medially, until the anterosuperior iliac spine laterally. In patients with bilateral hernia, two meshes were placed, one on each side respectively, surpassing the midline. The mesh was fixed with tuckers made of resorbable material (Securetrap®) or unabsorbable material (Protack®) according to the preference of the surgeon in charge of the procedure. The peritoneum was closed with continuous suture of slow absorbable material (Vycril®) or slow reabsorbed barb suture (Stratafix®). Local infiltration of all wounds was performed with ropivacaine at a dose of 3 mg / kg.

Surgical time was recorded as intraoperative variables, which was defined as minutes from the preparation of the surgical site to the closure of the skin; the type of hernia according to Nyhus classification and the presence of intraoperative complications.

At the end of the procedure, the patients were transferred to the recovery room. During the postoperative recovery an analgesic scheme was stipulated according to need. The rescues were made according to the evaluation of the nurse and the treating anesthetist and consisted of the following levels:

* First level: ketorolac 30 mg EV or diclofenac 75 mg EV. In patients with decreased glomerular filtration, paracetamol 1000 mg EV was used.
* Second level: morphine 1 - 3 mg EV. When the requirements of the ambulatory surgery guide of the Asociación Argentina de Cirugía listed in table N° 1 were fulfilled, the patient was discharged from hospital. The same was in charge of the responsible surgeon, who delivered the postoperative indications verbally and in writing, confirming the understanding of them by the patient and the companion.

The length of stay in the unit was recorded, as well as the need to administer analgesics during the same and pain according to the visual analog scale (EVA) at discharge.

Feasibility is expressed as the percentage of patients who were referred from the outpatient surgery unit.

The data about postoperative complications were collected prospectively through ambulatory controls previously stipulated at 7, 30, 180 and 360 days. They are classified into early (up to 30 days of the procedure) and late. The first included seroma, surgical site infection and hematoma; and late trocar hernias, recurrence and postoperative pain. Chronic postoperative pain is one that persists beyond the third month after the procedure.

In the first ambulatory control consultation at 7 days, patients were asked to rate their level of satisfaction with the procedure by choosing one of the four categories: not satisfied, not very satisfied, satisfied and very satisfied For the study of costs in addition to outpatients, those patients who underwent laparoscopic inguinal hernia in the inpatient setting during the period analyzed were included in the analysis. In this way, two branches of study were drawn up, one corresponding to patients operated on an outpatient basis and the other to patients operated through a hospital regimen.

Being a surgical procedure performed under a different hospital regime, a cost minimization study was carried out taking the average cost of performing an ambulatory procedure versus the same requiring admission.

When considering the economic situation of the República Argentina in the time under study (devaluation of the peso argentino weight of 100% and inflation of approximately 30% per year), continuous patients operated between December 2016 and April 2017 were taken, which represents the average of the period under study, as representative samples of each branch. For each patient, the surgical time, the persistence time in the ambulatory anesthetic recovery room or the hospitalization room, and the time of postoperative hospitalization were recorded in a database.

The materials used during surgery and anesthesia were previously standardized so that all the patients who underwent this procedure used the same resources.

The cost department of the Hospital Italiano de Buenos Aires was responsible for collecting the costs of each of these patients. They were divided into fixed costs per procedure, per hour/operating room, per hour in the ambulatory surgery recovery room, per hour in the recovery room of the central operating room and per day of hospitalization.

The costs were calculated in Argentine Pesos (AP) and converted into US Dollars (USD) taking into account the exchange rate in January 2017: 1 USD = 16.30 PA.

The categorical data were described as percentages and the quantitative data as mean and standard deviation or median and interquartile range according to the observed distribution. To compare means of quantitative variables, Student's t-test or Mann-Whitney U test was used according to the observed distribution. Chi-square or Fisher's test was used for the rest of the variables. A p <.05 was considered significant.

Regression models were constructed to adjust for confounding potentials.

ELIGIBILITY:
1. Inclusion Criteria:

   * Patients older than 18 years old
   * Laparoscopic inguinal hernioplasty as the pincipal surgery
2. Exclusion Criteria:

   * Patients with, high anesthetic risk (decompensated ASA III and ASA IV)
   * Morbid obesity (higher BMI 40),
   * Sleep apnea with indication of use of CPAP (Continuous Positive Airway Pressure)
   * Medicated psychiatric disease,
   * Drug-dependent patient
   * Patients with an inadequate social environment-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 with no major comorbidities that required a laparoscopic inguinal hernioplasty
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Incidence of surgical Complications | Patients follow up is 12 month
  Incidence of seroma, Incidence of hematoma, % of reoperation, incidence of wound infection
Costs of the procedure | One month after surgery
  Cost of laparoscopic hernioplasty in ambulatory surgery center. Cost of laparoscopic hernioplasty when required hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Scaravonati, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Ciudad de Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided
I have not decided yet. Maybe some data could be share to other researchers

REFERENCES:
- [Background] Jenkins JT, O'Dwyer PJ. Inguinal hernias. BMJ. 2008 Feb 2;336(7638):269-72. doi: 10.1136/bmj.39450.428275.AD. No abstract available. PMID 18244999
- [Background] Neumayer L, Giobbie-Hurder A, Jonasson O, Fitzgibbons R Jr, Dunlop D, Gibbs J, Reda D, Henderson W; Veterans Affairs Cooperative Studies Program 456 Investigators. Open mesh versus laparoscopic mesh repair of inguinal hernia. N Engl J Med. 2004 Apr 29;350(18):1819-27. doi: 10.1056/NEJMoa040093. Epub 2004 Apr 25. PMID 15107485
- [Background] Payne JH Jr, Grininger LM, Izawa MT, Podoll EF, Lindahl PJ, Balfour J. Laparoscopic or open inguinal herniorrhaphy? A randomized prospective trial. Arch Surg. 1994 Sep;129(9):973-9; discussion 979-81. doi: 10.1001/archsurg.1994.01420330087016. PMID 8080380
- [Background] Simons MP, Aufenacker T, Bay-Nielsen M, Bouillot JL, Campanelli G, Conze J, de Lange D, Fortelny R, Heikkinen T, Kingsnorth A, Kukleta J, Morales-Conde S, Nordin P, Schumpelick V, Smedberg S, Smietanski M, Weber G, Miserez M. European Hernia Society guidelines on the treatment of inguinal hernia in adult patients. Hernia. 2009 Aug;13(4):343-403. doi: 10.1007/s10029-009-0529-7. Epub 2009 Jul 28. PMID 19636493
- [Background] Miserez M, Peeters E, Aufenacker T, Bouillot JL, Campanelli G, Conze J, Fortelny R, Heikkinen T, Jorgensen LN, Kukleta J, Morales-Conde S, Nordin P, Schumpelick V, Smedberg S, Smietanski M, Weber G, Simons MP. Update with level 1 studies of the European Hernia Society guidelines on the treatment of inguinal hernia in adult patients. Hernia. 2014 Apr;18(2):151-63. doi: 10.1007/s10029-014-1236-6. Epub 2014 Mar 20. PMID 24647885
- [Background] McCloud JM, Evans DS. Day-case laparoscopic hernia repair in a single unit. Surg Endosc. 2003 Mar;17(3):491-3. doi: 10.1007/s00464-002-9093-2. Epub 2002 Nov 6. PMID 12415338